CLINICAL TRIAL: NCT06064500
Title: A Phase 3b, Multicenter, Single-arm, Expanded Access Protocol of Tarlatamab (AMG 757) for the Treatment of Subjects With Advanced Small Cell Lung Cancer After Two or More Prior Lines of Treatment
Brief Title: Tarlatamab (AMG 757) Expanded Access Protocol for Advanced Small Cell Lung Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20220100
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Small Cell Lung Cancer
Keywords: Lung cancer; Extensive-stage small cell lung cancer; Tarlatamab; AMG 757; Bispecific T-Cell Engager; BiTE; Immunotherapy; Immuno-oncology; Delta-like ligand 3
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms; Bites and Stings | interventions — AMG 757

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered as a 60-minute intravenous infusion with 1 mg step dose on cycle 1 day 1 followed by a 10 mg target dose on cycle 1 day 8 and cycle 1 day 15 in a 28-day cycle. Subsequent doses (10 mg) will be administered every 2 weeks.
  Other Names: AMG 757

SUMMARY:
The primary objective of the study is to provide expanded access to and characterize the safety profile of tarlatamab in participants with advanced small cell lung cancer (SCLC) after two or more prior lines of treatment (including at least one platinum-based regimen).

EA may still be available in countries outside of the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed SCLC
* Extensive-stage, unable to be encompassed in a tolerable radiation plan
* Progressed or recurred following 1 platinum-based regimen and at least 1 other prior line of therapy
* Eastern Cooperative Oncology Group (ECOG) PS of 0 to 1
* Minimum life expectancy of 12 weeks

Exclusion Criteria:

* Any previous diagnosis of transformed non-small cell lung cancer (NSCLC), epidermal growth factor receptor (EGFR) activating mutation positive NSCLC that has transformed to SCLC, or mixed SCLC NSCLC histology
* Symptomatic central nervous system (CNS) metastases
* Active hepatitis B or hepatitis C virus infection
* Eligible for participation in any Amgen-sponsored ongoing clinical study of the investigational product
* Currently or previously enrolled in a prior tarlatamab study
* Female participants and/or male participants with female partners who are pregnant, breastfeeding, planning to become pregnant or donate eggs while on study through 60 days after the last dose of tarlatamab
* Male and female participants unwilling to practice abstinence and/or use protocol specified method of contraception

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- United States (9):
  - Yale School of Medicine, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Martin Memorial Health System, Stuart, Florida
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Perlmutter Cancer Center at New York University Langone Hospital - 34th Street, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Cancer Care Northwest - South, Spokane, Washington
- Brazil (2):
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
- Israel (4):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital-Ein Kerem, Jerusalem
  - Assuta Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
- Japan (8):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com